CLINICAL TRIAL: NCT01685073
Title: The Role of Sleep in the Treatment of Cannabis Use Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00068969; U01DA031784 (NIH)
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Drug Addiction
Keywords: marijuana; cannabis; treatment; insomnia; relapse
MeSH Terms: conditions — Substance-Related Disorders; Marijuana Abuse; Sleep Initiation and Maintenance Disorders; Recurrence | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zolpidem (Experimental): Participants receive active zolpidem nightly in addition to psychosocial therapy during 12-week treatment of a cannabis use disorder
  Interventions: Drug: Zolpidem extended-release; Behavioral: MET/CBT
- Placebo (Placebo Comparator): Participants receive placebo medication during a 12-week psychosocial treatment for a cannabis use disorder
  Interventions: Behavioral: MET/CBT

INTERVENTIONS:
Drug: Zolpidem extended-release — nightly administration of zolpidem extended-release
  Other Names: Ambien CR
  Arms: Zolpidem
Behavioral: MET/CBT — a standardized 12-week therapy consisting of motivational enhancement therapy (MET) and cognitive behavior therapy (CBT) for treating cannabis use disorders will be administered to all study participants

SUMMARY:
The number of people seeking treatment for marijuana-related problems is on the rise, yet there is no currently accepted medication proven to help them quit. Frequent marijuana users have reported that they have trouble sleeping when they try to quit, and that the loss of sleep can lead to relapse. This research is designed to measure the severity of sleep problems in people as they are trying to quit heavy use of marijuana, and to investigate whether extended-release zolpidem (Ambien CR®) can improve quit rates among people trying to stop using marijuana.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 years.
2. Recent problematic use of cannabis
3. Cannabis use impacts sleep

Exclusion Criteria:

1. Dependent on drugs other than cannabis or nicotine, or current Axis I psychiatric disorder
2. Moderate sleep apnea or periodic limb movement disorder
3. Pregnant, breast feeding, or planning to become pregnant within the next 3 months
4. Current condition associated with severe cognitive/social impairment
5. Allergy to any ingredient in extended-release zolpidem or prior adverse reaction to zolpidem
6. Current use of drugs that affect metabolism via cytochrome P450 or current illness resulting in severe hepatic impairment
7. Current use of hypnotic medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2012-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pacek LR, Herrmann ES, Smith MT, Vandrey R. Sleep continuity, architecture and quality among treatment-seeking cannabis users: An in-home, unattended polysomnographic study. Exp Clin Psychopharmacol. 2017 Aug;25(4):295-302. doi: 10.1037/pha0000126. PMID 28782982

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zolpidem | Placebo
Started | 62 (Randomized) | 65 (Randomized)
Completed | 32 (Retained in treatment through 12 weeks) | 33 (Retained in treatment through 12 weeks)
Not Completed | 30 | 32
Not completed — Lost to Follow-up | 6 | 8
Not completed — Withdrawal by Subject | 24 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zolpidem | Placebo | Total
Number analyzed (Participants) | 62 | 65 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (9) | 32 (9) | 31 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 37 | 42 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 57 | 63 | 120
  Unknown or Not Reported | 0 | 0 | 0
Tobacco Smoking Status [Count of Participants; unit: Participants] — Tobacco smoking status count was for participants who answered YES to tobacco smoking
  Participants | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency as Assessed by Percentage of Time Asleep While in Bed
Description: Percentage of time asleep while in bed is measured using ambulatory polysomnography (PSG) equipment.
Time Frame: Week 1 of treatment
Population: Sleep data was not obtained for 12 people in the zolpidem group and 14 people in the placebo group at Week 1, and could not be included in this analysis. These individuals dropped out of the study or were lost to follow-up by the time of data collection.
Measure: Mean (Standard Deviation); unit: percentage of time asleep while in bed
Arm/Group | Zolpidem | Placebo
Number analyzed (Participants) | 50 | 51
percentage of time asleep while in bed | 78 (16) | 74 (19)

2. Primary Outcome: Number of Participants With Cannabis Abstinence as Assessed by Urine Cannabis Testing
Description: Qualitative urine cannabis testing outcomes of study participants; missing drop-outs presumed positive; Negative = THCCOOH <50ng/mL via EIA.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Zolpidem | Placebo
Number analyzed (Participants) | 62 | 65
Participants
  Negative urine test | 17 | 10
  Positive urine test | 45 | 55

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Zolpidem | Placebo
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/65
Serious Adverse Events (participants affected / at risk) | 2/62 | 0/65
Other Adverse Events (participants affected / at risk) | 30/62 | 35/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolpidem (N=62) | Placebo (N=65)
Stroke, cerebrovascular accident (Vascular disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolpidem (N=62) | Placebo (N=65)
toothache (General disorders) | 5 (5) | 3 (3)
Headache (General disorders) | 4 (4) | 5 (5)
Cold symptoms (General disorders) | 6 (6) | 9 (9)
nausea (Gastrointestinal disorders) | 7 (7) | 7 (7)
emesis (Gastrointestinal disorders) | 6 (6) | 6 (6)
Sleep Difficulties (General disorders) | 2 (2) | 5 (5)

LIMITATIONS AND CAVEATS:
There was a significant number of participant drop-outs in both study arms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT01685073/Prot_SAP_000.pdf